CLINICAL TRIAL: NCT05781217
Title: Short Versus Long-term Androgen Deprivation Therapy Combined With Salvage Radiotherapy in Prostate Cancer Patients With Biochemical Recurrence After Prostatectomy: a Multicentre Phase III Randomised Controlled Trial
Brief Title: Short Versus Long-term Androgen Deprivation Therapy With Salvage Radiotherapy in Prostate Cancer. URONCOR 0624
Acronym: URONCOR 06-24
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Investigación en Oncología Radioterápica - Fundación Española de Oncología Radioterápic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URONCOR 06-24
Record Dates: First submitted 2023-02-24; First posted 2023-03-23 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer; Salvage Radiotherapy; Biochemical Recurrence; Androgen Deprivation Therapy; Metastases-free Survival
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triptorelin Pamoate; Goserelin; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- short-term ADT (6 months) (Active Comparator): ARM 1:
  LHRH analogues for 6 months + bicalutamide 50 for 30 days
  Interventions: Drug: triptorelin, goserelin, leuprorelin
- long-term ADT (24 months) (Active Comparator): LHRH analogues for 24 months + bicalutamide 50 for 30 days
  Interventions: Drug: triptorelin, goserelin, leuprorelin

INTERVENTIONS:
Drug: triptorelin, goserelin, leuprorelin — ADT will consist of LHRH analogues (triptorelin, goserelin, leuprorelin) with bicalutamide 50 mg/day started 10 days before the first ADT injection to avoid LHRH-related flare-ups. Bicalutamide will be discontinued after 30 days. The LHRH analogue will be initiated prior to the start of radiotherapy and administered for 6 or 24 months depending on treatment allocation. The maximum time permitted between randomisation and administration of the first LHRH dose is 30 days. The maximum time from the first LHRH dose to the start of SRT is 60 days.

SUMMARY:
The optimal indication for ADT has long been a point of controversy, at least until the results of randomised trials comparing RT with and without ADT were published. NCCN guidelines and most retrospective series and left the decision to prescribe ADT in combination with RT to the discretion of the treating physician, despite a lack of clear scientific evidence to support this recommendation. The percentage of patients in those retrospective series who received hormone therapy ranged from 33% to 71%, but generally involved patients with adverse prognostic factors (Gleason score > 7, stage pT3-T4, PSA > 1 ng/mL in cases with biochemical recurrence [BCR], and PSA doubling time [PSA-DT] < 6 months). Despite the heterogeneity in those studies in terms of treatment duration, RT dose, and treatment volumes, most of the studies found that ADT significantly prolonged biochemical relapse-free survival (BRFS), especially in patients with PSA levels > 1 ng/mL at recurrence.

The results of two randomised trials evaluating SRT with or without ADT were published in 2017, with both trials demonstrating a benefit for ADT in this clinical setting. A follow-up study confirmed the value of ADT in combination with SRT in terms of better PFS and, in the RTOG study, an improvement in overall survival (OS). Despite the lack of data from phase III trials regarding the influence of PSA-DT, the BRFS interval, and the Gleason score in terms of their effects on the clinical course of patients who develop BCR, there is strong evidence from other studies to support the use of these variables (together with age and comorbidities). Given the available evidence, we believe that these variables should be considered when determining the indications for ADT.

In line with the philosophy underlying the approach used by D'Amico to develop a risk classification system for prostate cancer patients at diagnosis, we propose three risk groups. According to Pollack et al. and Spratt et al., low-risk patients would not benefit from hormone therapy, especially long-term ADT, due to the deleterious effects of such treatment. By contrast, intermediate and high risk patients would be candidates for ADT combined with RT. However, the optimal duration of ADT in these patients (6 months vs. 2 years) remains undefined and needs to be determined prospectively in a randomised trial, similar to the approach used in the DART 05.01 trial.

SRT and ADT are widely used in routine clinical practice to treat patients who develop BCR after prostatectomy. In this context, we intend to perform a multicentre, phase III trial to define the optimal duration of ADT (6 vs. 24 months).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically-confirmed prostate cancer treated with radical prostatectomy. Patients who have not undergone lymph node dissection are eligible for inclusion.
2. Biochemical recurrence after prostatectomy: BCR is defined as a PSA value ≥ 0.2 ng/mL, with at least one confirmatory PSA determination ≥ two weeks after the first test (the confirmatory PSA level must be higher than the initial value). Patients with Gleason 8-10, pT3b or R1 are eligible for inclusion in the trial with PSA ≥ 0.15 ng/mL; however, in patients with PSA > 0.4 ng/mL, imaging tests (conventional CT and bone scans or advanced imaging techniques such as PSMA or choline PET/CT) should be performed to check for metastases. In patients with PSA levels between 0.15 and 0.4 ng/mL, no further tests are required to check for distant metastases prior to inclusion.
3. Intermediate and high-risk patients according to the classification criteria proposed by González San Segundo et al. (18):

   CHARACTERISTICS INTERMEDIATE RISK (≥ 2) HIGH RISK(≥ 1)

   PSA at diagnosis, ng/mL 0.6-1.0 ≥1.0 PSA doubling time, months 6-12 < 6 GLEASON / ISUP 7/3 ≥8/≥4 TNM (prostatectomy specimen) pT2-3a pN0-Mx pT3b pN0-Mx Time to biochemical recurrence, months >18 <18 Margins Positive Positive
4. Testosterone level > 150 ng/dL at inclusion
5. ECOG 0-1
6. Life expectancy > 5 years
7. Signed informed consent

Exclusion Criteria:

1. Presence of pN1 disease in the original surgical specimen
2. Presence of macroscopic disease on imaging tests. If the PSA at diagnosis is > 0.4 ng/mL, then imaging tests (CT and bone scan and/or PET/CT or body magnetic resonance imaging [MRI]) are required.
3. PSA <0.2 or <0.15 ng/mL (if Gleason score=10, pT3b, or R1 in the radical prostatectomy specimen).
4. Previous pelvic radiotherapy
5. Radiotherapy contraindicated
6. Ongoing treatment with ADT or PSA-modulating drugs (e.g., finasteride, dutasteride, high dose steroids)
7. Inability to understand the treatment protocol or sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
To compare 5-year MFS rates in prostate cancer patients treated with long- versus short-term ADT in combination with salvage radiotherapy | 5 years
  Distant metastasis-free survival: time from administration of the first LHRH analogue (this same starting point applies to all secondary objectives) until the patient develops M1a disease (involved retroperitoneal lymph nodes) or M1b-c disease (bone/visceral involvement) according to RECIST 1.1 criteria based on conventional computed tomography (CT) imaging and bone scans. The use of advanced molecular imaging-PSMA or choline positron-emission tomography (PET)/CT-is subject to the centre-specific protocols in place at the participating hospitals; however, metastatic progression will be determined according to RECIST 1.1 criteria based on conventional imaging tests.

SECONDARY OUTCOMES:
To compare the two study arms in terms of the Biochemical-relapse free interval | 5 years
  BRFS: time to biochemical progression defined as an increase in PSA confirmed by a second PSA determination (0.2 ng/mL above the salvage radiotherapy nadir or a sustained elevation in PSA levels).
To compare the two study arms in terms of the Pelvic progression-free survival | 5 years
  Pelvic PFS: time to local recurrence (prostate bed) and/or N1 disease (positive lymph nodes below the aortic bifurcation) according to RECIST 1.1 criteria by conventional CT imaging and bone scan. The use of advanced molecular imaging (PSMA or choline PET/CT) will depend on centre-specific protocols; determination of metastatic progression will be based on RECIST 1.1 criteria from conventional imaging tests.
To compare the two study arms in terms of the Time to start of cytotoxic treatment | 5 years
  Cytotoxic treatment-free interval: time to the start of the first cytotoxic treatment or local treatment for oligorecurrence.
To compare the two study arms in terms of the Time to castration resistance | 5 years
  Time interval to castration resistance: the time to biochemical and/or clinical progression with castration levels (testosterone < 50 ng/dL). Progression to castration resistance is defined as three consecutive increases in PSA (one-week intervals) with at least two PSA increases > 2 ng/mL and a 50% increase over the PSA nadir, progression of bone lesions (≥ two lesions on the bone scan), progression of soft tissue lesions (RECIST 1.1 criteria), or the development of ≥ one soft tissue or visceral metastases (including lymph nodes).
To compare the two study arms in terms of the Cancer-specific survival | 5 years
  time to death due to prostate cancer or treatment-related complications
To compare the two study arms in terms of the Overall survival | 5 years
  time to death from any cause
To compare the two study arms in terms of the Acute and late toxicity | 5 years
  Acute toxicity: toxicity (CTCAE criteria, v. 4.0; https://evs.nci.nih.gov) appearing any time from treatment initiation up to three months after completion of RT.
To compare the two study arms in terms of the Late toxicity | 5 years
  -Late toxicity: from 3 months to 5 years after completing RT (CTCAE v 4.0).
To compare the two study arms in terms of Quality of life (QoL) | 5 years
  Quality of life (QoL): from baseline (prior to RT) to five years after completion of RT, assessed with the EORTC QLQ-C30 and QLQ-PR25 questionnaires.

CONTACTS AND LOCATIONS:
Locations (17):
- Spain (17):
  - Instituto Catalán de Oncología Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Quirón Madrid, Pozuelo de Alarcón, Madrid
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital San Francisco de Asís, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario de La Paz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Sant Joan de Reus, Tarragona
  - Hospital Universitario y Politécnico de La Fe, Valencia

REFERENCES:
- [Background] Parker CC, Clarke NW, Cook AD, Kynaston HG, Petersen PM, Catton C, Cross W, Logue J, Parulekar W, Payne H, Persad R, Pickering H, Saad F, Anderson J, Bahl A, Bottomley D, Brasso K, Chahal R, Cooke PW, Eddy B, Gibbs S, Goh C, Gujral S, Heath C, Henderson A, Jaganathan R, Jakobsen H, James ND, Kanaga Sundaram S, Lees K, Lester J, Lindberg H, Money-Kyrle J, Morris S, O'Sullivan J, Ostler P, Owen L, Patel P, Pope A, Popert R, Raman R, Roder MA, Sayers I, Simms M, Wilson J, Zarkar A, Parmar MKB, Sydes MR. Timing of radiotherapy after radical prostatectomy (RADICALS-RT): a randomised, controlled phase 3 trial. Lancet. 2020 Oct 31;396(10260):1413-1421. doi: 10.1016/S0140-6736(20)31553-1. Epub 2020 Sep 28. PMID 33002429
- [Background] Sargos P, Chabaud S, Latorzeff I, Magne N, Benyoucef A, Supiot S, Pasquier D, Abdiche MS, Gilliot O, Graff-Cailleaud P, Silva M, Bergerot P, Baumann P, Belkacemi Y, Azria D, Brihoum M, Soulie M, Richaud P. Adjuvant radiotherapy versus early salvage radiotherapy plus short-term androgen deprivation therapy in men with localised prostate cancer after radical prostatectomy (GETUG-AFU 17): a randomised, phase 3 trial. Lancet Oncol. 2020 Oct;21(10):1341-1352. doi: 10.1016/S1470-2045(20)30454-X. PMID 33002438
- [Background] Kneebone A, Fraser-Browne C, Duchesne GM, Fisher R, Frydenberg M, Herschtal A, Williams SG, Brown C, Delprado W, Haworth A, Joseph DJ, Martin JM, Matthews JHL, Millar JL, Sidhom M, Spry N, Tang CI, Turner S, Wiltshire KL, Woo HH, Davis ID, Lim TS, Pearse M. Adjuvant radiotherapy versus early salvage radiotherapy following radical prostatectomy (TROG 08.03/ANZUP RAVES): a randomised, controlled, phase 3, non-inferiority trial. Lancet Oncol. 2020 Oct;21(10):1331-1340. doi: 10.1016/S1470-2045(20)30456-3. PMID 33002437
- [Background] Vale CL, Fisher D, Kneebone A, Parker C, Pearse M, Richaud P, Sargos P, Sydes MR, Brawley C, Brihoum M, Brown C, Chabaud S, Cook A, Forcat S, Fraser-Browne C, Latorzeff I, Parmar MKB, Tierney JF; ARTISTIC Meta-analysis Group. Adjuvant or early salvage radiotherapy for the treatment of localised and locally advanced prostate cancer: a prospectively planned systematic review and meta-analysis of aggregate data. Lancet. 2020 Oct 31;396(10260):1422-1431. doi: 10.1016/S0140-6736(20)31952-8. Epub 2020 Sep 28. PMID 33002431
- [Background] Lieng H, Hayden AJ, Christie DRH, Davis BJ, Eade TN, Emmett L, Holt T, Hruby G, Pryor D, Shakespeare TP, Sidhom M, Skala M, Wiltshire K, Yaxley J, Kneebone A. Radiotherapy for recurrent prostate cancer: 2018 Recommendations of the Australian and New Zealand Radiation Oncology Genito-Urinary group. Radiother Oncol. 2018 Nov;129(2):377-386. doi: 10.1016/j.radonc.2018.06.027. Epub 2018 Jul 20. PMID 30037499
- [Background] Shipley WU, Seiferheld W, Lukka HR, Major PP, Heney NM, Grignon DJ, Sartor O, Patel MP, Bahary JP, Zietman AL, Pisansky TM, Zeitzer KL, Lawton CA, Feng FY, Lovett RD, Balogh AG, Souhami L, Rosenthal SA, Kerlin KJ, Dignam JJ, Pugh SL, Sandler HM; NRG Oncology RTOG. Radiation with or without Antiandrogen Therapy in Recurrent Prostate Cancer. N Engl J Med. 2017 Feb 2;376(5):417-428. doi: 10.1056/NEJMoa1607529. PMID 28146658
- [Background] Carrie C, Hasbini A, de Laroche G, Richaud P, Guerif S, Latorzeff I, Supiot S, Bosset M, Lagrange JL, Beckendorf V, Lesaunier F, Dubray B, Wagner JP, N'Guyen TD, Suchaud JP, Crehange G, Barbier N, Habibian M, Ferlay C, Fourneret P, Ruffion A, Dussart S. Salvage radiotherapy with or without short-term hormone therapy for rising prostate-specific antigen concentration after radical prostatectomy (GETUG-AFU 16): a randomised, multicentre, open-label phase 3 trial. Lancet Oncol. 2016 Jun;17(6):747-756. doi: 10.1016/S1470-2045(16)00111-X. Epub 2016 May 6. PMID 27160475
- [Background] Valicenti RK, Thompson I Jr, Albertsen P, Davis BJ, Goldenberg SL, Wolf JS, Sartor O, Klein E, Hahn C, Michalski J, Roach M 3rd, Faraday MM; American Society for Radiation Oncology/American Urological Association. Adjuvant and salvage radiation therapy after prostatectomy: American Society for Radiation Oncology/American Urological Association guidelines. Int J Radiat Oncol Biol Phys. 2013 Aug 1;86(5):822-8. doi: 10.1016/j.ijrobp.2013.05.029. PMID 23845839
- [Background] Fossati N, Karnes RJ, Boorjian SA, Moschini M, Morlacco A, Bossi A, Seisen T, Cozzarini C, Fiorino C, Noris Chiorda B, Gandaglia G, Dell'Oglio P, Joniau S, Tosco L, Shariat S, Goldner G, Hinkelbein W, Bartkowiak D, Haustermans K, Tombal B, Montorsi F, Van Poppel H, Wiegel T, Briganti A. Long-term Impact of Adjuvant Versus Early Salvage Radiation Therapy in pT3N0 Prostate Cancer Patients Treated with Radical Prostatectomy: Results from a Multi-institutional Series. Eur Urol. 2017 Jun;71(6):886-893. doi: 10.1016/j.eururo.2016.07.028. Epub 2016 Jul 30. PMID 27484843
- [Background] Spratt DE, Dess RT, Zumsteg ZS, Lin DW, Tran PT, Morgan TM, Antonarakis ES, Nguyen PL, Ryan CJ, Sandler HM, Cooperberg MR, Posadas E, Feng FY. A Systematic Review and Framework for the Use of Hormone Therapy with Salvage Radiation Therapy for Recurrent Prostate Cancer. Eur Urol. 2018 Feb;73(2):156-165. doi: 10.1016/j.eururo.2017.06.027. Epub 2017 Jul 14. PMID 28716370
- [Background] Gonzalez-San Segundo C, Counago F, Gomez-Iturriaga A. Androgen Deprivation Therapy and Salvage Radiotherapy: Are We Missing Something? Eur Urol. 2019 Aug;76(2):260-261. doi: 10.1016/j.eururo.2019.01.045. Epub 2019 Feb 8. No abstract available. PMID 30745145
- [Background] Jia ZW, Chang K, Dai B, Kong YY, Wang Y, Qu YY, Zhu YP, Ye DW. Factors influencing biochemical recurrence in patients who have received salvage radiotherapy after radical prostatectomy: a systematic review and meta-analysis. Asian J Androl. 2017 Jul-Aug;19(4):493-499. doi: 10.4103/1008-682X.179531. PMID 27241314
- [Background] Carrie C, Magne N, Burban-Provost P, Sargos P, Latorzeff I, Lagrange JL, Supiot S, Belkacemi Y, Peiffert D, Allouache N, Dubray BM, Servagi-Vernat S, Suchaud JP, Crehange G, Guerif S, Brihoum M, Barbier N, Graff-Cailleaud P, Ruffion A, Dussart S, Ferlay C, Chabaud S. Short-term androgen deprivation therapy combined with radiotherapy as salvage treatment after radical prostatectomy for prostate cancer (GETUG-AFU 16): a 112-month follow-up of a phase 3, randomised trial. Lancet Oncol. 2019 Dec;20(12):1740-1749. doi: 10.1016/S1470-2045(19)30486-3. Epub 2019 Oct 16. PMID 31629656
- [Background] Dess RT, Sun Y, Jackson WC, Jairath NK, Kishan AU, Wallington DG, Mahal BA, Stish BJ, Zumsteg ZS, Den RB, Hall WA, Gharzai LA, Jaworski EM, Reichert ZR, Morgan TM, Mehra R, Schaeffer EM, Sartor O, Nguyen PL, Lee WR, Rosenthal SA, Michalski JM, Schipper MJ, Dignam JJ, Pisansky TM, Zietman AL, Sandler HM, Efstathiou JA, Feng FY, Shipley WU, Spratt DE. Association of Presalvage Radiotherapy PSA Levels After Prostatectomy With Outcomes of Long-term Antiandrogen Therapy in Men With Prostate Cancer. JAMA Oncol. 2020 May 1;6(5):735-743. doi: 10.1001/jamaoncol.2020.0109. PMID 32215583
- [Background] Pollack A, Karrison TG, Balogh AG, Gomella LG, Low DA, Bruner DW, Wefel JS, Martin AG, Michalski JM, Angyalfi SJ, Lukka H, Faria SL, Rodrigues GB, Beauchemin MC, Lee RJ, Seaward SA, Allen AM, Monitto DC, Seiferheld W, Sartor O, Feng F, Sandler HM. The addition of androgen deprivation therapy and pelvic lymph node treatment to prostate bed salvage radiotherapy (NRG Oncology/RTOG 0534 SPPORT): an international, multicentre, randomised phase 3 trial. Lancet. 2022 May 14;399(10338):1886-1901. doi: 10.1016/S0140-6736(21)01790-6. PMID 35569466
- [Background] Yokomizo A, Wakabayashi M, Satoh T, Hashine K, Inoue T, Fujimoto K, Egawa S, Habuchi T, Kawashima K, Ishizuka O, Shinohara N, Sugimoto M, Yoshino Y, Nihei K, Fukuda H, Tobisu KI, Kakehi Y, Naito S; JCOG0401 Investigators. Salvage Radiotherapy Versus Hormone Therapy for Prostate-specific Antigen Failure After Radical Prostatectomy: A Randomised, Multicentre, Open-label, Phase 3 Trial (JCOG0401)dagger. Eur Urol. 2020 Jun;77(6):689-698. doi: 10.1016/j.eururo.2019.11.023. Epub 2019 Dec 19. PMID 31866092
- [Background] Van den Broeck T, van den Bergh RCN, Arfi N, Gross T, Moris L, Briers E, Cumberbatch M, De Santis M, Tilki D, Fanti S, Fossati N, Gillessen S, Grummet JP, Henry AM, Lardas M, Liew M, Rouviere O, Pecanka J, Mason MD, Schoots IG, van Der Kwast TH, van Der Poel HG, Wiegel T, Willemse PM, Yuan Y, Lam TB, Cornford P, Mottet N. Prognostic Value of Biochemical Recurrence Following Treatment with Curative Intent for Prostate Cancer: A Systematic Review. Eur Urol. 2019 Jun;75(6):967-987. doi: 10.1016/j.eururo.2018.10.011. Epub 2018 Oct 17. PMID 30342843
- [Background] Zapatero A, Guerrero A, Maldonado X, Alvarez A, San-Segundo CG, Rodriguez MAC, Sole JM, Olive AP, Casas F, Boladeras A, de Vidales CM, de la Torre MLV, Vara S, Sanz JL, Calvo FA. High-dose radiotherapy and risk-adapted androgen deprivation in localised prostate cancer (DART 01/05): 10-year results of a phase 3 randomised, controlled trial. Lancet Oncol. 2022 May;23(5):671-681. doi: 10.1016/S1470-2045(22)00190-5. Epub 2022 Apr 12. PMID 35427469
- [Background] Poortmans P, Bossi A, Vandeputte K, Bosset M, Miralbell R, Maingon P, Boehmer D, Budiharto T, Symon Z, van den Bergh AC, Scrase C, Van Poppel H, Bolla M; EORTC Radiation Oncology Group. Guidelines for target volume definition in post-operative radiotherapy for prostate cancer, on behalf of the EORTC Radiation Oncology Group. Radiother Oncol. 2007 Aug;84(2):121-7. doi: 10.1016/j.radonc.2007.07.017. Epub 2007 Aug 13. PMID 17706307
- [Background] Michalski JM, Lawton C, El Naqa I, Ritter M, O'Meara E, Seider MJ, Lee WR, Rosenthal SA, Pisansky T, Catton C, Valicenti RK, Zietman AL, Bosch WR, Sandler H, Buyyounouski MK, Menard C. Development of RTOG consensus guidelines for the definition of the clinical target volume for postoperative conformal radiation therapy for prostate cancer. Int J Radiat Oncol Biol Phys. 2010 Feb 1;76(2):361-8. doi: 10.1016/j.ijrobp.2009.02.006. Epub 2009 Apr 23. PMID 19394158
- [Background] Robin S, Jolicoeur M, Palumbo S, Zilli T, Crehange G, De Hertogh O, Derashodian T, Sargos P, Salembier C, Supiot S, Udrescu C, Chapet O. Prostate Bed Delineation Guidelines for Postoperative Radiation Therapy: On Behalf Of The Francophone Group of Urological Radiation Therapy. Int J Radiat Oncol Biol Phys. 2021 Apr 1;109(5):1243-1253. doi: 10.1016/j.ijrobp.2020.11.010. Epub 2020 Nov 10. PMID 33186618
- [Background] Sidhom MA, Kneebone AB, Lehman M, Wiltshire KL, Millar JL, Mukherjee RK, Shakespeare TP, Tai KH. Post-prostatectomy radiation therapy: consensus guidelines of the Australian and New Zealand Radiation Oncology Genito-Urinary Group. Radiother Oncol. 2008 Jul;88(1):10-9. doi: 10.1016/j.radonc.2008.05.006. Epub 2008 May 29. PMID 18514340
- [Background] Fossati N, Robesti D, Karnes RJ, Soligo M, Boorjian SA, Bossi A, Coraggio G, Di Muzio N, Cozzarini C, Noris Chiorda B, Gandaglia G, Scarcella S, Bartkowiak D, Bohmer D, Shariat S, Goldner G, Battaglia A, Joniau S, Haustermans K, De Meerleer G, Fonteyne V, Ost P, Van Poppel H, Montorsi F, Wiegel T, Briganti A. Assessing the Role and Optimal Duration of Hormonal Treatment in Association with Salvage Radiation Therapy After Radical Prostatectomy: Results from a Multi-Institutional Study. Eur Urol. 2019 Oct;76(4):443-449. doi: 10.1016/j.eururo.2019.02.004. Epub 2019 Feb 22. PMID 30799187
- [Background] Jackson WC, Schipper MJ, Johnson SB, Foster C, Li D, Sandler HM, Palapattu GS, Hamstra DA, Feng FY. Duration of Androgen Deprivation Therapy Influences Outcomes for Patients Receiving Radiation Therapy Following Radical Prostatectomy. Eur Urol. 2016 Jan;69(1):50-7. doi: 10.1016/j.eururo.2015.05.009. Epub 2015 May 21. PMID 26004800
- [Derived] Gonzalez-San Segundo C, Lopez Campos F, Gomez Iturriaga A, Rodriguez A, Olivera J, Duque-Santana V, Sancho G, Henriquez I, Conde AJ, Valero J, Maldonado X, Glaria L, Caballero B, Sanmamed N, Mases J, Boladeras-Inglada AM, Montijano M, Santos M, Alvarez A, Martinez JI, Counago F. A randomised trial of short- vs long-term androgen deprivation with salvage radiotherapy for biochemical failure following radical prostatectomy: URONCOR 06-24. BJU Int. 2024 Oct;134(4):568-577. doi: 10.1111/bju.16484. Epub 2024 Jul 23. PMID 39041411